CLINICAL TRIAL: NCT06052540
Title: Effetto Della Supplementazione di Una Miscela di Ceppi Probiotici (Bifidobacterium Breve M-16V, Bifidobacterium Lactis HN019, Lactobacillus Rhamnosus HN001) in Bambini Febbrili Con Infezioni Delle Alte Vie Respiratorie
Brief Title: Probiotic Supplementation in Children Affected by Upper Respiratory Infections
Acronym: PROBIOS2021
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Principal Investigator, Cristiana Berti, Researcher, Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 726_2021bis
Record Dates: First submitted 2023-09-19; First posted 2023-09-25 (Actual); Last update posted 2023-09-29 (Actual); Status verified 2023-09

CONDITIONS: Upper Respiratory Tract Infection
Keywords: probiotic; children; respiratory infection
MeSH Terms: conditions — Respiratory Tract Infections

STUDY DESIGN:
Who Masked: Participant, Investigator, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Probiotics (Active Comparator): Probiotic supplement: Mix of probiotic strails. Administration: 1 stick per day or 5 drops per day. Study duration for each patient: 14 days.
  Interventions: Dietary Supplement: Probiotic supplement
- Placebo (Placebo Comparator): Placebo: Medium Chain Triglycerides. Administration: 1 stick per day or 5 drops per day. Study duration for each patient: 14 days.
  Interventions: Dietary Supplement: Placebo

INTERVENTIONS:
Dietary Supplement: Probiotic supplement — * Stick: Bifidobacterium breve M-16V, Bifidobacterium lactis HN019, Lactobacillus rhamnosus HN001 + Maltodestrins
  * Drops: Bifidobacterium breve M-16V, Bifidobacterium lactis HN019, Lactobacillus rhamnosus HN001 + Medium chain triglycerides, vegetable fats, emulsifier, and maltodextrin.
  Other Names: Ofmom SynterAct BIMBI
  Arms: Probiotics
Dietary Supplement: Placebo — * Drops: Medium Chain Triglycerides, vegetal oil, E471, and maltodextrin
  * Stick: Maltodextrin.
  Arms: Placebo

SUMMARY:
The goal of this randomized non-pharmacological Intervention study is to evaluate the effects of probiotic supplements (Bifidobacterium breve M-16V, Bifidobacterium lactis HN019, Lactobacillus rhamnosus HN001) on children affected by upper respiratory tract infections.

The main questions it aims to answer are:

* probiotic formulation can reduce intensity and duration of fever in children affected by upper respiratory tract infections
* probiotic formulation can influence the gut microbiota composition in children affected by upper respiratory tract infections

Participants will be asked to take probiotic supplements or placebo for 14 days and to collect three fecal samples: before probiotic supplementation (T0), 14 days after probiotic supplementation (T1), and 12 months after the enrollment (T2).

ELIGIBILITY:
Inclusion Criteria:

* Access to the Emergency room with fever and upper respiratory tract infection
* Age > 28 days and ≤ 4 years
* Signature of informed consent by parents or guardian

Exclusion Criteria:

* Presence of pathologies associated with immunosuppression or ongoing immunosuppressant treatments
* Hospitalisation/hospitalisation
* Diarrhea at enrollment
* No signed informed consent

Ages: 29 Days to 4 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 128 (Actual)
Dates: Start 2021-09-01 (Actual); Primary Completion 2023-06-30 (Actual); Study Completion 2024-06-30 (Estimated)

PRIMARY OUTCOMES:
Mean duration of fever in days by measuring body temperature | Approximatively 7 days
  To assess the effects of a probiotic supplement compaerd to a placebo on mean duration and intensity of fever measured by a thermometer

SECONDARY OUTCOMES:
Mean change in gut microbial composition by measuring gut microbiota characterization in fecal samples | 1 year
  To assess the effects of a probiotic supplement compared to a placebo on gut microbiota characteristics at baseline, 14 days and 12 months by generation Sequencing, real-time PCR, and typing PCR
Gastrointestinal symptoms | Approximatively 7 days
  Evaluation of the gastrointestinal symptoms by interview
Adverse events | Approximatively 15 days
  Evaluation of differences in clinical effects in subjects with or without antibiotics collected by interview

CONTACTS AND LOCATIONS:
Overall Officials: Carlo V Agostoni, Prof, Principal Investigator — Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milano, Italy
Locations (1):
- Fondazione IRCCS Ca' Granda Ospedale Maggiore Policlinico, Milan, Italy

REFERENCES:
- [Derived] Bettocchi S, Comotti A, Elli M, De Cosmi V, Berti C, Alberti I, Mazzocchi A, Rosazza C, Agostoni C, Milani GP. Probiotics and Fever Duration in Children With Upper Respiratory Tract Infections: A Randomized Clinical Trial. JAMA Netw Open. 2025 Mar 3;8(3):e250669. doi: 10.1001/jamanetworkopen.2025.0669. PMID 40085083